CLINICAL TRIAL: NCT07372729
Title: A Smart Wearable Devices-based Comprehensive Intervention Through a Cluster Randomized Controlled Trial to Improve Cardiovascular Health in Overweight/Obese Individuals With Cardiometabolic Preconditions
Brief Title: Smartwatch-based Intervention for Cardiovascular Health (SWITCH)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Cangzhou Central Hospital (Other); Health Community Group of Yuhuan People's Hosptial (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BJAZH-SWITCH-2026
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prehypertension; Borderline Dyslipidemia; Overweight , Obesity; Prediabetes
MeSH Terms: conditions — Prehypertension; Overweight; Obesity; Prediabetic State | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartwatch-Based Comprehensive Intervention (Experimental): Participants receive mHealth-based multi-faceted behavioral intervention via a closed-loop management pathway formed by the intervention tools of "smartwatch - mobile phone - data interaction and processing center - WeChat mini-program (WMP)".
  Interventions: Behavioral: Smartwatch-Based Multi-Faceted Behavioral Intervention Model Led by Exercise and Dietary Interventions, Supported by Primary Medical Staff, Along with the Distribution of Health Education Manuals
- Usual Care (Active Comparator): Participants in the control group will receive only face-to-face health education sessions.
  Interventions: Behavioral: Face-to-face health education sessions

INTERVENTIONS:
Behavioral: Smartwatch-Based Multi-Faceted Behavioral Intervention Model Led by Exercise and Dietary Interventions, Supported by Primary Medical Staff, Along with the Distribution of Health Education Manuals — The intervention model integrates multiple functions including data collection, intelligent analysis, and personalized intervention, and delivers targeted management for the target population. Among these, the intervention content includes the smartwatch-based comprehensive behavioral intervention model adopted in the model construction phase; for overweight/obese individuals with cardiometabolic preconditions, a customized combination of implementation strategies is provided. Intervention measures include smartwatch-based indicator monitoring and risk warning, diet and exercise reporting, monitoring, and goal setting/planning, community interaction, collaborative management by medical staff and family members.In addition, routine health education will be provided during face-to-face visits at baseline, 3 months, and 6 months.
  Arms: Smartwatch-Based Comprehensive Intervention
Behavioral: Face-to-face health education sessions — At baseline, 3 months, and 6 months, participants will attend follow-up visits at primary healthcare institutions in the project areas and receive usual care based on guideline-recommended health education manuals, which provide comprehensive lifestyle intervention advice.
  Arms: Usual Care

SUMMARY:
This study aims to employ a cluster randomized controlled trial to evaluate the effectiveness of an mHealth-Based Multi-faceted Cardiovascular Health Intervention Model among Overweight/Obese Individuals with Cardiometabolic Preconditions, thereby providing theoretical foundations and practical guidance for the prevention and management of this population.

DETAILED DESCRIPTION:
This study plans to evaluate the effectiveness of an mHealth-Based Multi-faceted Cardiovascular Health Intervention Model among Overweight/Obese Individuals with Cardiometabolic Preconditions through a cluster randomized controlled trial. The study is designed as a prospective, multicenter, parallel-group, open-label cluster randomized controlled trial. The objective is to compare the effects of a comprehensive behavioral intervention model versus usual care on improving cardiovascular health among community-dwelling individuals who are overweight/obese and have at least one of the following conditions: prehypertension, prediabetes, or borderline dyslipidemia. The trial plans to include approximately 40 clusters across three regions (covering both urban and rural areas), with an expected recruitment of more than 35 eligible participants per cluster, resulting in a total sample size of around 1,400 participants. Participants in the intervention group will receive a comprehensive behavioral intervention during the intensive phase (first 6 months), led by smartwatches and a WeChat mini-program (WMP), supported by primary healthcare providers and an integrated management platform, along with face-to-face health education. During the maintenance phase (subsequent 6 months), they will receive only self-management support via smartwatches and the , supplemented by face-to-face health education. Participants in the control group will receive only face-to-face health education throughout the study period. All participants will undergo follow-up assessments at 3, 6 and 12 months from baseline. The primary outcome is the change in Life's Essential 8 components (diet, physical activity, smoking, sleep, BMI, blood lipids, blood glucose, and blood pressure) at 6 months of intervention. Secondary outcomes include changes in the primary outcome at 12 months and improvements in each component of Life's Essential 8.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years, no gender restriction;
2. Overweight and obesity: Body Mass Index (BMI) 24.0-32.4 kg/m^2, or waist circumference >= 90 cm for males and >= 85 cm for females;
3. Presence of at least one metabolic high-risk state among prehypertension, prediabetes, or borderline elevated blood lipids, and without a diagnosis of hypertension, diabetes mellitus, or dyslipidemia:

(1) Prehypertension: Systolic blood pressure (SBP) 130-139 mmHg and/or diastolic blood pressure (DBP) 80-89 mmHg, without regular use of antihypertensive medication in the past month; (2) Prediabetes: Fasting blood glucose (FBG) 6.1-6.9 mmol/L, or glycated hemoglobin (HbA1c) 5.7%-6.4%, without regular use of hypoglycemic medication in the past month; (3) Borderline elevated blood lipids: Total cholesterol (TC) 5.2-6.1 mmol/L, or low-density lipoprotein cholesterol (LDL-C) 3.4-4.0 mmol/L, or triglycerides (TG) 1.7-2.2 mmol/L, or non-high-density lipoprotein cholesterol (non-HDL-C) 4.1-4.8 mmol/L, without regular use of lipid-lowering medication in the past month; 4. Local permanent residents who will reside in the area for at least 12 month after enrollment; 5. Have basic reading, writing, and comprehension abilities; proficient in using internet-connected smartphones; able to independently complete basic operations of the application; 6. Written informed consent provided.

Exclusion Criteria:

1. Secondary obesity diagnosed by doctors in secondary or higher-level medical institutions;
2. Cardiovascular and cerebrovascular diseases, including myocardial infarction, stroke, heart failure, arrhythmia; or having received coronary intervention therapy, cardiac surgery, etc.; or with a 10-year high risk of cardiovascular disease;
3. Diseases seriously affecting survival, such as malignant tumors, AIDS, hepatic and renal failure;
4. Pregnancy, lactation period, or women who may become pregnant within one year;
5. History of severe neuropsychiatric diseases with potential cognitive or communication impairments, such as dementia, Alzheimer's disease, Parkinson's syndrome;
6. Individuals with limited daily mobility;
7. Individuals undergoing or planning to receive weight loss through surgery, medication, or other methods;
8. Currently participating in other lifestyle intervention-related trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Life's Essential 8 risk score | Baseline and 6 months after intervention
  The primary outcome is change in Life's Essential 8 risk score from baseline and 6 months following intervention.
  The Life's Essential 8 (LE8) is a cardiovascular health score that uses a 0-100 scale. The score is calculated based on a participant's adherence to eight healthy lifestyle components: diet, physical activity, smoking habits, body mass index, non-HDL cholesterol, blood sugar, blood pressure, and sleep. Each component has scoring algorithm ranging from 0 to 100 points, allowing generation of a composite cardiovascular health score (the unweighted average of all components) that also varies from 0 to 100 points. 0 will indicate the lowest cardiovascular health scores and 100 will indicate the highest cardiovascular health scores.

SECONDARY OUTCOMES:
Blood pressure (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8 (LE8), including changes in blood pressure (both systolic and diastolic), will be assessed at baseline, 3 months, 6 months, and 12 months. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: <120/<80 mm Hg; 0 points: ≥160 mm Hg or ≥100 mm Hg.
non-HDL cholesterol(Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in non-HDL cholesterol, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: <3.36 mmol/L; 0 points: ≥5.69 mmol/L.
Blood glucose (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in blood glucose, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: No history of diabetes and hemoglobin A1c <5.7%; 0 points: Diabetes with hemoglobin A1c ≥10.0%
Body Mass Index (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in body mass index, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: <23 kg/m²; 0 points: ≥35 kg/m².
Physical activity (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in physical activity, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC).
  For the primary outcome composite score: 100 points: ≥150 minutes of moderate or vigorous activities per week; 0 points: 0 minutes.
Sleep (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in sleep, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: 7-<9 hours of sleep per night; 0 points: <4 hours of sleep per night.
Smoking habits (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in smoking habits, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: Never smoker; 0 points: Current smoker.
Health diet pattern (Individual Life's Essential 8 components) | Baseline and 3 months after intervention; Baseline and 6 months after intervention; Baseline and 12 months after intervention
  Changes in the individual risk factors of Life's Essential 8, including changes in diet patterns, will be assessed at baseline, 3 months, 6 months, and 12 months after intervention. Data will be derived from the Electronic Data Capture (EDC) system.
  For the primary outcome composite score: 100 points: DASH diet score of 8; 0 points: DASH diet score of 0 to 1.
Change in Life's Essential 8 risk score | Baseline and 3 months after intervention; Baseline and 12 months after intervention
  the change in the Life's Essential 8 risk score from baseline to 3 months and 12 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: yue qi, PhD, Principal Investigator — Beijing Anzhen Hospital

IPD SHARING:
Plan to Share IPD: No